CLINICAL TRIAL: NCT00116857
Title: Omega-3 for Depression and Other Cardiac Risk Factors
Brief Title: Omega-3 Fatty Acids to Improve Depression and Reduce Cardiovascular Risk Factors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Carney, Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 186; R01HL076808 (NIH)
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Results first posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Cardiovascular Diseases; Depression; Heart Diseases; Myocardial Infarction; Angina, Unstable
MeSH Terms: conditions — Cardiovascular Diseases; Depression; Heart Diseases; Myocardial Infarction; Angina, Unstable | interventions — Sertraline; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sertraline/omega-3 supplement (Active Comparator)
  Interventions: Drug: Sertraline/omega-3
- Sertraline/corn oil (Placebo Comparator)
  Interventions: Drug: Sertraline/Corn Oil

INTERVENTIONS:
Drug: Sertraline/omega-3 — Sertraline (50 mgs) plus omega-3 (2 grams)
  Arms: Sertraline/omega-3 supplement
Drug: Sertraline/Corn Oil — Sertraline (50 mgs) plus corn oil (2 grams) (placebo)
  Arms: Sertraline/corn oil

SUMMARY:
This study will determine the effects of omega-3 fatty acid (FA) augmentation of sertraline on depression and cardiac endpoints after myocardial infarction (MI).

DETAILED DESCRIPTION:
BACKGROUND:

Depression is a risk factor for morbidity and mortality following an acute MI and unstable angina. Two recent studies (sertraline versus placebo and sertraline plus cognitive therapy versus usual care) reported only modest reductions in depression following an acute MI or unstable angina, and many treated patients remained depressed. Neither study reported better medical outcomes in the treated patients. Earlier studies found that even subclinical depression increases the risk of mortality in cardiac patients. Thus, more effective treatments are needed to eliminate depression and improve medical outcomes in patients following an acute MI or unstable angina. Omega-3 FAs have been shown to augment the efficacy of antidepressants for major depression and to improve several cardiac risk factors. However, these findings have been shown in separate lines of research. No previous study has investigated whether omega-3 FAs can simultaneously improve depression and reduce cardiovascular risk factors in post-MI patients.

DESIGN NARRATIVE:

One hundred fifty patients who meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for a current major depressive episode and who score 15 or higher on the Beck Depression Inventory II with a history of acute MI, unstable angina, or other cardiac event will be enrolled in a randomized, double-blind, placebo-controlled trial of omega-3 augmentation of sertraline. The participants will be randomly assigned to receive either sertraline plus omega-3 or sertraline plus placebo for 10 weeks. At baseline and again after ten weeks, the subjects will complete the following: 1) assessments of depression and psychosocial functioning; 2) 24-hour electrocardiogram monitoring for heart rate variability analysis; and 3) blood draws to measure procoagulant and proinflammatory markers, and plasma levels of sertraline and omega-3. If this study shows that omega-3 reduces depression and improves cardiovascular disease markers, there will be a basis for proposing a larger clinical trial to determine whether it can also improve survival after hospitalization for acute MI or unstable angina.

ELIGIBILITY:
Inclusion Criteria:

* Meets the DSM-IV criteria for a current major depressive episode
* Score of 15 or higher on the Beck Depression Inventory II
* History of acute myocardial infarction, unstable angina, or documented coronary disease

Exclusion Criteria:

* Physician or patient refusal
* Lives far away from study site
* Current alcohol or drug abuse
* Psychosis, dementia, or bipolar disorder
* Already taking Omega-3
* Medically ill or disabled such that patient is unable to participate
* Comorbid illness likely to be fatal within 1 year of study entry
* Seizure disorder or takes anticonvulsants
* Pregnant or breast feeding
* Liver or kidney disease
* Severe hypertriglyceridemia (greater than 400 mg/dL)
* Bleeding or clotting disorder
* Type 2 diabetes with a hemoglobin A1c (HbA1c) level greater than 10
* Taking lithium or monoamine oxidase inhibitor (MAO-I)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2005-02; Primary Completion 2009-06 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert M. Carney, PhD, Study Chair — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

REFERENCES:
- [Result] Carney RM, Freedland KE, Rubin EH, Rich MW, Steinmeyer BC, Harris WS. Omega-3 augmentation of sertraline in treatment of depression in patients with coronary heart disease: a randomized controlled trial. JAMA. 2009 Oct 21;302(15):1651-7. doi: 10.1001/jama.2009.1487. PMID 19843899
- [Derived] Appleton KM, Voyias PD, Sallis HM, Dawson S, Ness AR, Churchill R, Perry R. Omega-3 fatty acids for depression in adults. Cochrane Database Syst Rev. 2021 Nov 24;11(11):CD004692. doi: 10.1002/14651858.CD004692.pub5. PMID 34817851
- [Derived] Carney RM, Steinmeyer BC, Freedland KE, Rubin EH, Rich MW, Harris WS. Baseline blood levels of omega-3 and depression remission: a secondary analysis of data from a placebo-controlled trial of omega-3 supplements. J Clin Psychiatry. 2016 Feb;77(2):e138-43. doi: 10.4088/JCP.14m09660. PMID 26930527
- [Derived] Bot M, Carney RM, Freedland KE, Rubin EH, Rich MW, Steinmeyer BC, Mann DL. Inflammation and treatment response to sertraline in patients with coronary heart disease and comorbid major depression. J Psychosom Res. 2011 Jul;71(1):13-7. doi: 10.1016/j.jpsychores.2010.11.006. Epub 2011 Jan 15. PMID 21665007

RESULTS

PARTICIPANT FLOW:
Groups:
- Sertraline Plus Omega-3 Supplement: Sertraline 50mg 1 tablet by mouth everyday. Plus Omega-3 supplement capsules 2g by mouth everyday.
- Sertraline/Corn Oil: Sertraline 50mg 1 tablet by mouth everyday. Plus corn oil placebo capsules 2 g by mouth everyday.
Period: Overall Study
Arm/Group | Sertraline Plus Omega-3 Supplement | Sertraline/Corn Oil
Started | 62 | 60
Completed | 59 | 56
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Sertraline Plus Omega-3 Supplement: Sertaline 50mg tablets 1 by mouth everyday, plus Omega-3 supplement capsules 2g by mouth everyday.
- Sertraline/Corn Oil: Sertaline 50mg tablets 1 by mouth everyday, plus corn oil placebo capsules 2g by mouth everyday.
- Total: Total of all reporting groups
Arm/Group | Sertraline Plus Omega-3 Supplement | Sertraline/Corn Oil | Total
Number analyzed (Participants) | 62 | 60 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 48 | 98
  >=65 years | 12 | 12 | 24
Age Continuous [Mean (Standard Deviation); unit: years] | 58.1 (9.4) | 58.6 (8.5) | 58.4 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 19 | 41
  Male | 40 | 41 | 81
Region of Enrollment [Number; unit: participants]
  United States | 62 | 60 | 122

OUTCOME MEASURES:

1. Primary Outcome: Beck Depression Inventory-II
Description: Beck Depression Inventory-II scores on a scale of 0 to 63, minimum score equals 0 maximum score equals 63. Higher value represents a worse outcome. Baseline scores are compared to scores after treatment.
Time Frame: Measured at Baseline and 10 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline Plus Omega-3 Supplement | Sertraline/Corn Oil
Number analyzed (Participants) | 62 | 60
units on a scale | 16.1 (10.2) | 14.8 (9.7)

ADVERSE EVENTS:
Arm/Group | Sertraline Plus Omega-3 Supplement | Sertraline/Corn Oil
Serious Adverse Events (participants affected / at risk) | 0/62 | 0/60
Other Adverse Events (participants affected / at risk) | 0/62 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No